CLINICAL TRIAL: NCT00308503
Title: Efficacy and Safety of Eplivanserin 5mg/Day on Sleep Maintenance Insomnia: A 6 Week, Multicenter, Randomized, Double -Blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of Eplivanserin 5mg/Day on Sleep Maintenance Insomnia
Acronym: EPOCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6220
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Sleep Initiation and Maintenance Disorders; Insomnia
Keywords: Primary Insomnia; Sleep Maintenance Insomnia; Awakening
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — SR 46349B

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 5 mg/day
  Interventions: Drug: eplivanserin (SR46349)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eplivanserin (SR46349) — oral administration
  Arms: 1
Drug: placebo — oral administration
  Arms: 2

SUMMARY:
The aim of the study is to confirm the efficacy of eplivanserin 5mg/day on sleep maintenance of patients with primary insomnia using night polysomnography recordings over a 6-week treatment period corresponding to a stabilization of improvement of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for at least one month preceding the study visit.
* Disturbance of sleep maintenance:

  * Based on patient' s information:

    * Patient has spent at least 6.5 hours and not more than 9.0 hours, in bed, each night, over the preceding two weeks,
    * Patient must complain of at least one hour of wakefulness after sleep onset for at least 3 nights per week over the preceding month,
    * Patient must report impact on daytime functioning associated with sleep maintenance insomnia

Inclusion will be based on the nocturnal polysomnography (NPSG) recordings performed at the sleep laboratory during the two screening nights.

Exclusion Criteria:

* Females who are lactating or who are pregnant, or of childbearing potential not using an acceptable form of contraception
* Patients presenting with acute or chronic pain resulting in insomnia
* Patients with current psychiatric disturbances
* Body mass index > 32
* Evidence of any clinically significant, severe or unstable, acute or chronically progressive medical or surgical disorder, or any condition that may interfere with the absorption, metabolism, distribution or excretion of the study drug, or may affect patient safety
* Clinically significant and abnormal electrocardiogram (ECG) (including QTc B > 500ms),
* A positive test for hepatitis B (hepatitis B surface [HBs] antigens) or C (hepatitis C virus [HCV] antibodies)
* Positive qualitative urine drug screen at screening
* Consumption of xanthine-containing beverages (i.e. tea, coffee, or cola) comprising usually more than 5 cups or glasses per day
* Use of any over-the-counter or prescription sleep medication, or of any substance with psychotropic effects or properties known to affect sleep/wake, within one week or five half-lives (whichever is longer), prior to screening
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month
* Based on medical history and/or NPSG:

  * primary hypersomnia
  * narcolepsy
  * breathing-related sleep disorder (apnea-hypopnea index > 10/hour of sleep)
  * circadian rhythm sleep disorder
  * parasomnia (e.g. somnambulism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline of night polysomnography Wake Time After Sleep Onset (PSG WASO) | week 6

SECONDARY OUTCOMES:
Change from baseline in general productivity domain of the FOSQ (Functional Outcome of Sleep Questionnaire) | week 6
Change from baseline in patient reported wake after sleep onset (pr-WASO) | week 6

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis, Bridgewater, New York, United States
- Sanofi-Aventis, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis, Laval, Canada